CLINICAL TRIAL: NCT02074904
Title: Brain Mechanisms of Topiramate's Effects on Heavy Drinking
Brief Title: Topiramate's Effects on Heavy Drinking
Acronym: TOPMRI
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: We terminated the study to run it as a sub-study of NCT02371889, which is a 13 week, placebo controlled, double-blind, trial of topiramate in heavy drinkers.
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TOP MRI
Record Dates: First submitted 2014-02-20; First posted 2014-02-28 (Estimated); Results first posted 2017-12-11 (Actual); Last update posted 2018-09-21 (Actual); Status verified 2017-12

CONDITIONS: Alcohol Drinking
MeSH Terms: conditions — Alcohol Drinking | interventions — Topiramate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Topiramate (Experimental): up to 200mg/day orally (over 8 weeks during which the dosage is gradually increased up to 200 mg orally and then maintained, and 1 week of medication taper)
  Interventions: Drug: Topiramate
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Topiramate
  Other Names: Topamax
  Arms: Topiramate
Drug: Placebo
  Arms: Placebo

SUMMARY:
The proposed project will utilize perfusion functional magnetic resonance imaging (fMRI) to examine the effects of topiramate on brain and behavioral responses in heavy drinkers to appetitive alcohol reminders (cues that motivate continued alcohol use and relapse). This project will yield novel findings on brain and behavioral responses to alcohol cues, the effects of topiramate on alcohol cue reactivity, and the mechanisms underlying topiramate's ability to blunt alcohol cue reactivity and heavy drinking.

DETAILED DESCRIPTION:
This project is a double-blind, randomized, placebo-controlled study of topiramate's effects on brain and behavior responses in heavy drinkers. Eligible volunteers who meet study criteria will be randomized to receive either topiramate or placebo with weekly visits and medication management sessions. Participants will complete two magnetic resonance imaging sessions. The first scan session will occur prior to starting study drug, and the second scan will occur following six weeks of study drug. This project will yield novel findings on brain and behavioral responses to alcohol cues, the effects of topiramate on alcohol cue reactivity, and the mechanisms underlying topiramate's ability to blunt alcohol cue reactivity and heavy drinking.

ELIGIBILITY:
Inclusion Criteria:

* Physically healthy, as determined by a comprehensive physical examination and approval of the study physician, males or females who drink alcohol, ages 18-60.
* Average weekly ethanol consumption of >24 standard drinks for men, or >18 standard drinks for women.
* Females must be non-pregnant, non-lactating and either be of non-childbearing potential (i.e. sterilized via hysterectomy or bilateral tubal ligation or at least 2 years postmenopausal) or of child bearing potential but practicing a medically acceptable method of birth control. Examples of medically acceptable methods for this protocol include: the birth control pill, intrauterine device, injection of Depo-Provera, Norplant, contraceptive patch, contraceptive ring, double-barrier methods (such as condoms and diaphragm/spermicide), male partner sterilization, abstinence (and agreement to continue abstinence or to use an acceptable method of contraception, as listed above, should sexual activity commence), and tubal ligation.
* Provide voluntary informed consent.
* Must be able to read. [Subjects are required to be able to read because there are several self-administered measures that they must read, understand and provide written answers.]
* Intelligence quotient of ≥ 80.

Exclusion Criteria:

* Current, clinically significant physical disease or abnormality on the basis of medical history, physical examination, or routine laboratory evaluation.
* History of head trauma or injury causing loss of consciousness, lasting more than five (5) minutes or associated with skull fracture or inter-cranial bleeding or abnormal MRI.
* Current major DSM-IV Axis I diagnoses other than alcohol use disorder (except nicotine use disorder).
* Presence of magnetically active irremovable prosthetics, plates, pins, permanent retainer, bullets, etc. (unless a radiologist confirms that it's presence is unproblematic). An x-ray may be obtained to determine eligibility given the possibility of a foreign body.
* History of a serious psychiatric illness including psychosis, bipolar disorder, or suicidal or homicidal intent.
* Current treatment with carbonic anhydrase inhibitors.
* Claustrophobia or other medical condition preventing subject from lying in the MRI for approximately one (1) hour.
* Current regular treatment with psychotropic medications (e.g., benzodiazepines, antidepressants), which affect neurotransmitter systems or a medication being used to treat alcohol use disorders (e.g., naltrexone, acamprosate).
* Vision problems that cannot be corrected with glasses.
* Body Mass Index (BMI) greater than or equal to 34, body girth greater than 52 inches and a head girth greater than 25 inches.
* History of stroke and/or stroke related spasticity.
* History of glaucoma or kidney stones.
* HIV positive.
* History of seizures.
* History of topiramate treatment for alcohol use disorder and report no treatment response.
* Current DSM-5 diagnosis of alcohol use disorder that is clinically too severe to permit them to participate in a research trial in which the goal is to stop or reduce drinking.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2015-05; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reagan R Wetherill, PhD, Principal Investigator — University of Pennsylvania; Henry R Kranzler, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Center for Studies of Addiction, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Topiramate: up to 200mg/day orally (over 8 weeks during which the dosage is gradually increased up to 200 mg orally and then maintained, and 1 week of medication taper)
  Topiramate
Period: Overall Study
Arm/Group | Topiramate | Placebo
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated to run as a sub-study of NCT02371889. No data will be entered due to privacy concerns.
Groups:
- Total: Total of all reporting groups
Arm/Group | Topiramate | Placebo | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Continuous
Sex: Female, Male
Race (NIH/OMB)
Region of Enrollment [unit: participants]
fMRI Response in the Ventral Striatum/Medial Orbitofrontal Cortex During Alcohol Cue Exposure

OUTCOME MEASURES:

1. Primary Outcome: fMRI Response in the Ventral Striatum/Medial Orbitofrontal Cortex During Alcohol Cue Exposure
Description: At baseline (prior to randomization), brain and behavioral responses will be significantly greater during alcohol cue exposure compared to non-alcohol cue exposure. Following 6 weeks of study drug, individuals receiving topiramate will demonstrate greater reductions in brain activity and drinking behavior compared to individuals receiving placebo. Individuals receiving placebo will exhibit responses similar to baseline responses.
Time Frame: baseline to after 6 weeks of study drug
Population: The study was terminated to run as a sub-study of NCT02371889. No data will be entered due to privacy concerns.
Arm/Group | Topiramate | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Drinking Days
Description: change in drinking days from baseline to 9 weeks
Time Frame: baseline and 9 weeks
Population: The study was terminated to run as a sub-study of NCT02371889. No data will be entered due to privacy concerns.
Arm/Group | Topiramate | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Gamma-glutamyl Transferase (GGT) or Carbohydrate-deficient Transferrin (CDT) Levels
Description: Change in gamma-glutamyl transferase (GGT) or carbohydrate-deficient transferrin (CDT) levels after 9 weeks of treatment.
Time Frame: baseline and Visit 9 (9 weeks)
Population: The study was terminated to run as a sub-study of NCT02371889. No data will be entered due to privacy concerns.
Arm/Group | Topiramate | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Heavy Drinking Days
Description: change in number of heavy drinking days from baseline to 9 weeks
Time Frame: baseline to 9 weeks
Population: The study was terminated to run as a sub-study of NCT02371889. No data will be entered due to privacy concerns.
Arm/Group | Topiramate | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Mean Alcohol Consumption
Description: change in mean alcohol consumption from baseline to 9 weeks
Time Frame: baseline to 9 weeks
Population: The study was terminated to run as a sub-study of NCT02371889. No data will be entered due to privacy concerns.
Arm/Group | Topiramate | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: The study was terminated to run as a sub-study of NCT02371889. There were no Adverse Events.
Arm/Group | Topiramate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

LIMITATIONS AND CAVEATS:
We terminated the study to run it as a sub-study of NCT02371889. We didn't enter results of the one subject randomized to study medication due to privacy concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-10): https://cdn.clinicaltrials.gov/large-docs/04/NCT02074904/Prot_SAP_000.pdf